CLINICAL TRIAL: NCT03749694
Title: Investigating Temporal Improvements in Survival Following ST-elevation Myocardial Infarction: A Causal Mediation Analysis Using the Myocardial Ischaemia National Audit Project, 2004-2013.
Brief Title: Investigating Temporal Improvements in Survival Following ST-elevation Myocardial Infarction.
Status: Completed | Type: Observational
Sponsor: University of Leeds (Other)
Responsible Party: Principal Investigator, Tatendashe Bernadette Dondo, Postdoctoral medical statistician, University of Leeds
Other Study IDs: PG/13/81/30474_STEMI
Record Dates: First submitted 2018-11-20; First posted 2018-11-21 (Actual); Last update posted 2018-11-21 (Actual); Status verified 2018-11

CONDITIONS: Acute Myocardial Infarction
Keywords: Acute Myocardial Infarction; mortality; evidence-based care; Myocardial Ischaemia National Audit Project; ST-elevation myocardial infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study was to use data from the Myocardial Ischaemia National Audit Project (MINAP) to investigate whether temporal improvements in survival were associated with changes in patients' baseline clinical risk or use of guideline-indicated treatments for the management of STEMI, and to determine the extent to which associations explained the temporal improvements in survival.

ELIGIBILITY:
Inclusion Criteria:

* aged 18 years or more
* patients hospitalised with ST-elevation myocardial infarction

Exclusion Criteria:

* patients hospitalised with phenotypes other than ST-elevation myocardial infarction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population comprised of 232,353 in hospital survivors of ST-elevation myocardial infarction recorded in the Myocardial Ischaemia National Audit Project registry between 2004 and June 2013.
Sampling Method: Non-Probability Sample
Enrollment: 232353 (Actual)
Dates: Start 2004-01-01 (Actual); Primary Completion 2013-06-30 (Actual); Study Completion 2013-06-30 (Actual)

PRIMARY OUTCOMES:
All cause mortality | one year

SECONDARY OUTCOMES:
All cause mortality | six months

CONTACTS AND LOCATIONS:
Overall Officials: Chris P Gale, FRCP, Principal Investigator — University of Leeds; Tatendashe B Dondo, PhD, Principal Investigator — University of Leeds; Marlous Hall, PhD, Principal Investigator — University of Leeds

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dondo TB, Hall M, Munyombwe T, Wilkinson C, Yadegarfar ME, Timmis A, Batin PD, Jernberg T, Fox KA, Gale CP. A nationwide causal mediation analysis of survival following ST-elevation myocardial infarction. Heart. 2020 May;106(10):765-771. doi: 10.1136/heartjnl-2019-315760. Epub 2019 Nov 15. PMID 31732655